CLINICAL TRIAL: NCT03460899
Title: Impact of Hypoglycaemia in Patients With Diabetes Mellitus Type 2 on Platelet Activation
Acronym: Diaplate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-2017-04
Record Dates: First submitted 2018-02-22; First posted 2018-03-09 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus With Hypoglycemia; Diabetes Mellitus, Type 2; Hypoglycemia; Hypoglycemic Episode
Keywords: Hypoglycaemia; Platelet activity; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clamp Arm (Experimental): All 14 subjects will undergo an Euglycaemic Clamp at Visit 2 as well as a Hyperinsulinaemic/Hypoglycaemic Clamp at Visit 3 with the Intervention of reaching certain plasma glucose levels for blood sampling regarding platelet activity parameters. Infusion of Dextrose and human soluble insulin (Actrapid) will be used to reach certain plasma glucose levels.
  Interventions: Other: Euglycaemic Clamp; Other: Hyperinsulinaemic/Hypoglycaemic Clamp

INTERVENTIONS:
Other: Euglycaemic Clamp — All 14 subjects will undergo an euglycaemic clamp at Visit 2 with a plasma Glucose target of 5.5 mmol/L +/- 10% (4 timepoints for platelet activity parameter blood sampling)
Other: Hyperinsulinaemic/Hypoglycaemic Clamp — All 14 subjects will undergo a hypoglycaemic/hyperinsulinaemic clamp at Visit 3 with 4 timepoints for platelet activity Parameter blood sampling 30 minutes after reaching certain plasma glucose plateaus (5.5 mmol/L; 3.5 mmol/L; 2.5 mmol/L; after recovery again at 5.5 mmol/L)

SUMMARY:
This experimental study is planned to investigate the impact of hypoglycaemia on platelet activation parameters (PAP) during a hyperinsulinaemic hypoglycaemic clamp study. The hypothesis that hypoglycaemia in patients with Diabetes Mellitus, Type 2 (T2DM) leads to increased platelet activation will be tested.

DETAILED DESCRIPTION:
Increased platelet activation is significantly involved in the pathophysiology of micro- and macrovascular diabetic complications. Previously performed studies suggested platelet activation in both, hyper- and hypoglycaemic states, leading to a potentially increased risk for thromboembolic complications. Hypoglycaemia, in particular severe hypoglycaemic episodes, has been associated with increased cardiovascular or overall mortality in previous studies. Potential mechanisms include arrhythmias or increased risk for thromboembolism, based on platelet activation and/or hypercoagulability.

The aim of this experimental study is to investigate the impact of hypoglycaemia on platelet activation parameters (PAP) during a hyperinsulinaemic hypoglycaemic clamp study. We hypothesize that Hypoglycaemia in patients with T2DM leads to increased platelet activation.

The primary objective is to investigate platelet activation during different levels of hypoglycaemia induced by a stepwise hyperinsulinaemic, hypoglycemic clamp experiment in patients with T2DM.

Active study duration will be 5 days for each study participant. 14 subjects with T2DM without history of cardiovascular events or manifest atherosclerosis will be enrolled. During this monocentric, single arm, open, mechanistic trial platelet activation and recovery at one week after the clamp experiment, changes of pro-atherothrombotic markers during the hypoglycaemic clamp as well as counter regulatory hormone response during the clamp will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-64 years (both inclusive) at the time of signing informed consent
* Subjects diagnosed with type 2 diabetes (diagnosed regarding world health organization [WHO] criteria) and on stable treatment for a period of 90 days prior to screening with metformin as monotherapy or diet only. Stable is defined as unchanged dose
* Body mass index (BMI) between 20.0 and 35.0 kg/m2 (both inclusive)
* HbA1c between 43 and 64 mmol/mol (6.0% - 8.0%) (both inclusive)
* No use of platelet inhibiting therapy (e.g. aspirin, clopidogrel, ticagrelor, prasugrel)

Exclusion Criteria:

* All other forms of diabetes (type 1 diabetes, gestational diabetes) than type 2 diabetes mellitus
* Treatment with any glucose lowering agent(s) other than metformin in a period of 60 days before screening. An exception is short-term treatment (≤ 7 days in total) with insulin due to intercurrent illness
* Impaired hypoglycaemic awareness determined at the discretion of the investigator
* Medical history of arrhythmia as atrial fibrillation, atrial flutter, atrioventricular dissociation disorders or ventricular arrhythmias
* Previously known cardiovascular disease and / or past cardiovascular events, or past episodes of a congestive heart failure syndrome (NYHA II - NYHA IV)
* Severe hypoglycaemic event requiring third party help in the last 6 months
* Known allergy to human insulin or dextrose solution
* Clinically significant abnormal haematology, biochemistry, lipids, hormones, coagulation or urinalysis
* Uncontrolled hypertension defined as resting blood pressure at screening (after resting for 5 min, measured in sitting position) outside the range of 90-160 mmHg for systolic or 50-100 mmHg for diastolic
* Chronic liver failure with severe liver dysfunction as assessed by the investigator
* Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) levels > 3x upper Limit of normal (ULN)
* estimated Glomerular Filtration Rate (eGFR) <45 ml/min/1,73 m2
* Any musculoskeletal disorders holding back from stay in bed in a lying position during the time of the clamp experiments
* Treatment with beta-blockers, antiarrhythmic agents or neuroleptic drugs
* Active smoker or intake of illicit substances
* Regular intake of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Any mental disorders or psychiatric conditions which may interfere with understanding or conduction of study related procedures
* Females of child bearing potential without adequate contraceptive methods (i.e. sterilisation, intrauterine device, vasectomised partner; or medical history of hysterectomy)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, Principal Investigator — Medical University of Graz, Division of Endocrinology and Diabetology
Locations (1):
- Medical University of Graz, Department for Internal Medicine, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eyileten C, Wicik Z, Keshwani D, Aziz F, Aberer F, Pferschy PN, Tripolt NJ, Sourij C, Prietl B, Pruller F, von Lewinski D, De Rosa S, Siller-Matula JM, Postula M, Sourij H. Alteration of circulating platelet-related and diabetes-related microRNAs in individuals with type 2 diabetes mellitus: a stepwise hypoglycaemic clamp study. Cardiovasc Diabetol. 2022 May 20;21(1):79. doi: 10.1186/s12933-022-01517-5. PMID 35596173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Approximately 3 Months (End of February until beginning of May 2018)
  Recruitmet process: Subjects were recruited by using a local recruitment registry.
Groups:
- Clamp Arm: All 14 subjects will undergo an Euglycaemic Clamp at Visit 2 as well as a Hyperinsulinaemic/Hypoglycaemic Clamp at Visit 3 with the Intervention of reaching certain plasma glucose levels for blood sampling regarding platelet activity parameters. Infusion of Dextrose and human soluble insuline (Actrapid) will be used to reach certain plasma glucose levels.
  Euglycaemic Clamp: All 14 subjects will undergo an euglycaemic clamp at Visit 2 with a plasma Glucose target of 5.5 mmol/L +/- 10% (4 timepoints for platelet activity parameter blood sampling)
  Hyperinsulinaemic/Hypoglycaemic Clamp: All 14 subjects will undergo a hypoglycaemic/hyperinsulinaemic clamp at Visit 3 with 4 timepoints for platelet activity Parameter blood sampling 30 minutes after reaching certain plasma glucose plateaus (5.5 mmol/L; 3.5 mmol/L; 2.5 mmol/L; after recovery again at 5.5 mmol/L)
Period: Euglycaemic Clamp
Arm/Group | Clamp Arm
Started | 14 (First Euglycaemic Clamp completed: 05. March 2018)
Completed | 14 (Last Euglycaemic clamp completed: 23. May 2018)
Not Completed | 0
Period: Hyperinsulinaemic/Hypoglycaemic Clamp
Arm/Group | Clamp Arm
Started | 14 (First Hyperinsulinaemic/Hypoglycaemic Clamp completed: 15. March 2018)
Completed | 14 (Last Hyperinsulinaemic/Hypoglycaemic Clamp completed: 05. June 2018)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clamp Arm
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 28.9 (3.3)
Weight [Mean (Standard Deviation); unit: kg] | 86.4 (15.1)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 133 (13)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 83 (8)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 7.2 (0.9)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.02 (1.33)
Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.22 (1.19)
High-density lipoprotein-cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] | 1.19 (0.36)
Low-density lipoprotein-cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] | 3.13 (1.01)
Diabetes duration [Mean (Standard Deviation); unit: years] | 5 (4)
Daily metformin dose [Mean (Standard Deviation); unit: mg] | 1336 (599)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 51 (7)
Angiotensin-converting-enzyme inhibitors [Count of Participants; unit: Participants] | 4
Angiotensin-II receptor antagonists [Count of Participants; unit: Participants] | 5
Calcium antagonists [Count of Participants; unit: Participants] | 3
Diuretics [Count of Participants; unit: Participants] | 1
Statins [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Changes in Platelet Activation Marker Adenosin Diphosphate (%)
Description: Changes in platelet activation measured by light transmittance aggregometry (LTA) on a Chronolog 700 Lumi-Aggregometer based on Adenosin Diphosphate (ADP %) activation.
  Visit 3, Hyperinsulinaemic/Hypoglycaemic clamp Experiment:
  Timepoint 0 (Baseline = Plasma Glucose 100mg/dL [5.5mmol/L]) Timepoint 1 (Hypoglycaemia Plateau 1 = Plasma Glucose 63mg/dL [3.5mmol/L]) Timepoint 2 (Hypoglycaemia Plateau 2 = Plasma Glucose 45mg/dL [2.5mmol/L]) Timepoint 3 (Recovery = Plasma Glucose 100mg/dL [5.5mmol/L]
  Follow up 1 (1 Day after the Clamp Experiment) Follow up 2 (7 +/- 1 day after the Clamp Experiment)
Time Frame: Measurement during different levels of hypoglycaemia as well as 1 and 7 days after the clamp experiment
Measure: Mean (Standard Deviation); unit: percentage of ADP
Arm/Group | Clamp Arm
Number analyzed (Participants) | 14
percentage of ADP
  Timepoint 0 | 63 (14.3)
  Timepoint 1 | 64.4 (16.7)
  Timepoint 2 | 64.4 (13.4)
  Timepoint 3 | 61.1 (15.1)
  Follow up 1 | 67.7 (11.3)
  Follow up 2 | 70.4 (7.3)

2. Secondary Outcome: Quantification of Platelet Function and Activation PAC1CD62PCD63POS (%)
Description: Quantification of platelet activation markers by flow cytometry in unstimulated blood samples (CD62P, CD63 and binding of PAC-1) using a BD LSRFortessa flow cytometer.
  Hyperinsulinaemic/Hypoglycaemic clamp Experiment:
  Timepoint 0 (Baseline = Plasma Glucose 100mg/dL [5.5mmol/L]) Timepoint 1 (Hypoglycaemia Plateau 1 = Plasma Glucose 63mg/dL [3.5mmol/L]) Timepoint 2 (Hypoglycaemia Plateau 2 = Plasma Glucose 45mg/dL [2.5mmol/L]) Timepoint 3 (Recovery = Plasma Glucose 100mg/dL [5.5mmol/L]
  Follow up 1 (1 Day after the Clamp Experiment) Follow up 2 (7 +/- 1 day after the Clamp Experiment)
Time Frame: Measurement during different levels of hypoglycaemia as well as 1 and 7 days after the clamp experiment
Measure: Mean (Standard Deviation); unit: percentage of PAC1CD62PCD63POS
Arm/Group | Clamp Arm
Number analyzed (Participants) | 14
percentage of PAC1CD62PCD63POS
  Timepoint 0 | 0.023 (0.019)
  Timepoint 1 | 0.027 (0.028)
  Timepoint 2 | 0.032 (0.032)
  Timepoint 3 | 0.031 (0.033)
  Follow up 1 | 0.085 (0.071)
  Follow up 2 | 0.094 (0.087)

3. Secondary Outcome: Markers of Coagulation Plasminogen Activator Inhibitor-1 (ng/mL)
Description: Effects on coagulation parameter plasminogen activator Inhibitor-1 (PAI-1) measured by Enzyme-linked immunosorbent assays.
  Visit 3, Hyperinsulinaemic/Hypoglycaemic clamp Experiment:
  Timepoint 0 (Baseline = PG 100mg/dL [5.5mmol/L]) Timepoint 1 (Hypoglycaemia Plateau 1 = PG 63mg/dL [3.5mmol/L]) Timepoint 2 (Hypoglycaemia Plateau 2 = PG 45mg/dL [2.5mmol/L]) Timepoint 3 (Recovery = PG 100mg/dL [5.5mmol/L]
  Follow up 1 (1 Day after the Clamp Experiment) Follow up 2 (7 +/- 1 day after the Clamp Experiment)
Time Frame: Measurement during different levels of hypoglycaemia as well as 1 and 7 days after the clamp experiment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Clamp Arm
Number analyzed (Participants) | 14
ng/mL
  Timepoint 0 | 14.14 (9.06)
  Timepoint 1 | 11.32 (7.69)
  Timepoint 2 | 12.08 (8.50)
  Timepoin 3 | 13.50 (9.87)
  Follow up 1 | 26.26 (15.14)
  Follow up 2 | 25.35 (14.38)

4. Secondary Outcome: Changes in Coagulation Marker Fibrinogen (g/L)
Description: Changes in coagulation marker Fibrinogen, measured on a Behring Coagulation System BCS XP Analyzer.
  Visit 3, Hyperinsulinaemic/Hypoglycaemic clamp Experiment:
  Timepoint 0 (Baseline = PG 100mg/dL [5.5mmol/L]) Timepoint 1 (Hypoglycaemia Plateau 1 = PG 63mg/dL [3.5mmol/L]) Timepoint 2 (Hypoglycaemia Plateau 2 = PG 45mg/dL [2.5mmol/L]) Timepoint 3 (Recovery = PG 100mg/dL [5.5mmol/L]
  Follow up 1 (1 Day after the Clamp Experiment) Follow up 2 (7 +/- 1 day after the Clamp Experiment)
Time Frame: Measurement during different levels of hypoglycaemia as well as 1 and 7 days after the clamp experiment
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Clamp Arm
Number analyzed (Participants) | 14
g/L
  Timepoint 0 | 2.49 (0.40)
  Timepoint 1 | 2.54 (0.43)
  Timepoint 2 | 2.64 (0.45)
  Timepoint 3 | 2.49 (0.41)
  Follow up 1 | 2.90 (0.50)
  Follow up 2 | 2.93 (0.53)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for Adverse Events from successful Screening until Visit 5 Minimum timeframe for AE assessment: 18 days Maximum timeframe for AE assessment: 42 days
Arm/Group | Clamp Arm
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clamp Arm (N=14)
Abdominal pain (Hepatobiliary disorders) | 1 (1) — Episode of abdominal pain due to known cholecystolithiasis with hospitalization

LIMITATIONS AND CAVEATS:
14 subjects could be considered a small patient Group. Given the delayed activation of platelet and coagulation markers in our study, we still can not answer the question, at which glycaemic threshold this activation occurs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03460899/Prot_SAP_001.pdf